CLINICAL TRIAL: NCT05307562
Title: Efficacy of Respiratory Rehabilitation After COVID-19 Severe Infection
Acronym: COVFIS2021
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Gerard Muñoz, Principal Investigator. PhD, PT, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVFIS2021
Record Dates: First submitted 2022-02-18; First posted 2022-04-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: COVID-19 Respiratory Infection; Rehabilitation; Physical Therapists
Keywords: covid-19; training program; respiratory physiotherapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training program (Active Comparator): Global intervallic exercise using cyclometer and analytical strength exercises
  Interventions: Other: Interval training + analytical strength
- Training program + Inspiratory muscle traioning (IMT) (Experimental): Global intervallic exercise using cyclometer and analytical strength exercises + inspiratory muscles training
  Interventions: Other: Interval training + analytical strength and IMT

INTERVENTIONS:
Other: Interval training + analytical strength — Patients will receive a training program
  Arms: Training program
Other: Interval training + analytical strength and IMT — Patients will receive a training program + IMT
  Arms: Training program + Inspiratory muscle traioning (IMT)

SUMMARY:
The purpose of this study is to investigate the effects of a training program in patients that have suffered a COVID infection

DETAILED DESCRIPTION:
Once patients have been selected and meet inclusion criteria, they will sign informed consent. They will make a first visit to obtain the basal parameters. Once done, they will start the individualized training program for 12 weeks 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years
* Patients discharged from the Pulmonology Service with a diagnosis of COVID-19 by positive PCR and with severe pneumonia.
* At least three months after the presence of at least one of the following criteria:

  1. MRC dyspnea greater than or equal to 2.
  2. Decrease in the meters walked with respect to the reference values in the 6-minute walking test.

     C) Decreased respiratory muscle strength measured at Maximum Inspiratory Pressure (PIM) and / or Maximum Expiratory Pressure (PEM) with respect to reference values.
* Sign informed consent from the study

Exclusion Criteria:

* Patients who do not want to be included in the study.
* Pregnant women.
* Impossibility to perform ergometry or ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
changes in walking distance in the 6 minutes walk test | Baseline and 12 weeks after
  6MWT is a submaximal test performed in 30 meters corridor.

SECONDARY OUTCOMES:
changes in the maximum watts generated | Baseline and 12 weeks after
  Cardiopulmonary exercise test will be performed as maximal test
changes in (oxygen consumption) VO2 max | Baseline and 12 weeks after
  Cardiopulmonary exercise test will be performed as maximal test
changes in peak VO2 | Baseline and 12 weeks after
  Cardiopulmonary exercise test will be performed as maximal test
changes in the diaphragmatic path | Baseline and 12 weeks after
  Diaphragm echocardiography will be performed
changes in diaphragm thickness | Baseline and 12 weeks after
  Diaphragm echocardiography will be performed
changes in diaphragmatic shortening | Baseline and 12 weeks after
  Diaphragm echocardiography will be performed
changes in dyspnea | Baseline and 12 weeks after
  Measured with mMRC scale (scores from 0-4)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Muñoz, PhD, Principal Investigator — Girona Biomedical Research Institute
Locations (1):
- Josep Trueta University Hospital, Girona, Spain